CLINICAL TRIAL: NCT05804058
Title: Assessment of Biofilm Composition as a Predictive Biomarker for Prosthetic Joint Infection
Brief Title: Biofilm Composition as a Predictive Biomarker for Prosthetic Joint Infection
Acronym: Biofilms
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: University of Portsmouth (Other)
Responsible Party: Sponsor
Other Study IDs: PHT/2019/31
Record Dates: First submitted 2019-08-16; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Joint Infection
MeSH Terms: interventions — Reoperation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Synovial Fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthopaedic Patients: Patients due to undergo prosthetic hip revision surgery
  Interventions: Procedure: Revision surgery

INTERVENTIONS:
Procedure: Revision surgery — Patients due to undergo prosthetic revision surgery for any reason (infection or aseptic)

SUMMARY:
Prosthetic joint infection (PJI) represents one of the most common reasons for failure among hip and knee prostheses, with an incidence of around 1-2%. Infection can occur early (within days of surgery) or late (over a year after surgery), and no specific early markers for infection onset exist. Given the significant costs to the NHS for corrective revision surgery, the added suffering and risk to patients from surgery, and the risk of enhancing antimicrobial resistance through the use of broad-spectrum antibiotics, a more specific predictive test for early onset of infection is required.

DETAILED DESCRIPTION:
Over 80% of human infection is estimated to be a result of biofilm formation. Biofilms are an accumulation of microorganisms (predominantly bacteria) on a surface, resulting in a functional community which provides antibiotic resistance and a beneficial environment for the growth of pathogenic species that would otherwise be removed by the body's defences.

The use of medical implants in modern medicine has become an increasingly common occurrence, with hip and knee arthroplasty accounting for a large number of medical implant surgeries. Unfortunately, infections frequently result in failure of the implanted device (around 1-2% for knee and hip arthroplasty), requiring extensive revision surgery. Currently, no predictive biomarkers for PJI exist, and diagnostic tests require infection to have already taken hold and may often be highly invasive. Research conducted by the NIH suggests that accumulation of bacteria (known as biofilms) may account for over 80% of microbial infections in the human body and have been shown to develop on medical implants, such as those used in hip and knee arthroplasty. Bacterial biofilms on medical implants are poorly understood, making treatment very complex.

The investigators aim to identify early predictive biomarkers for PJI based on assessment of the biofilm structure on implants removed in revision surgery, either as a result of PJI or due to aseptic causes such as mechanical failure. The investigators will explore biofilm formation on hip joint prostheses using next generation sequencing (NGS) and 3D phase-contrast X-ray microscopy, and will compare bacterial diversity and biofilm structure between infected and non-infected samples to answer three main questions:

1. Can The investigators accurately describe the characteristic microbiome of hip joint prosthetic biofilms?
2. Is there a distinct characteristic microbiome or biofilm structure associated with PJI?
3. Can The investigators detect such characteristic biofilm members as biomarkers in simple blood tests?

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or above.
* Due to undergo prosthetic revision surgery for any reason identified by the clinical team Willing to provide informed consent

Exclusion Criteria:

* Participant lacking capacity to give informed consent
* Any other clinical reason the participant should not be included in the study- at the discretion of the clinical team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with symptoms likely to require revision hip surgery for correction.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Characteristic Formation of bacterial biofilm on orthopaedic implants | 1 day study visit
  measured by infection assessment- this is the term for the measure

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No